CLINICAL TRIAL: NCT05011890
Title: Feasibility and Acceptability of Remote Monitoring of Lung Cancer Patient-Reported Outcomes Using Moovcare®
Brief Title: Remote Monitoring of Lung Cancer Patient-Reported Outcomes Using Moovcare®
Acronym: LC-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Sivan Innovation Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC 2050; 25210 (Other Grant/Funding Number: Sivan Innovation Ltd)
Record Dates: First submitted 2021-07-26; First posted 2021-08-18 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Lung Cancer; Neoplasms, Lung; Neoplasms, Pulmonary; Pulmonary Cancer; Pulmonary Neoplasms; Cancer of Lung
Keywords: Patient Reported Outcome; Feasibility; Acceptability; Moovcare®
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single site nonrandomized feasibility study, participants on treatment and/or surveillance for new or existing diagnoses of lung cancer were assigned to a single arm involving monitoring of their patient-reported outcomes using a mobile medical application. The study population will include patients with a diagnosis of lung cancer undergoing outpatient treatment or surveillance at UNC. Patients will be recruited from the Multidisciplinary Thoracic Oncology Program (MTOP) clinics at the University of North Carolina over 10-12 months and undergo ePRO monitoring for 6 months or until criteria for coming off study are met, whichever comes first.
Masking Description: This is a single site non-randomized feasibility study. Participants on treatment and/or surveillance for new or existing diagnoses of lung cancer were assigned to monitor their patient-reported outcomes using a mobile medical application. The study population includes patients with a diagnosis of lung cancer undergoing outpatient treatment or surveillance at UNC. Patients were recruited from the Multidisciplinary Thoracic Oncology Program clinics at the University of North Carolina over 10-12 months and undergo ePRO monitoring for 6 months or until criteria for coming off study are met, whichever comes first.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single-arm (Other): Participants will be assigned to the single-arm involving weekly monitoring of their patient-reported outcomes using Moovcare®.
  Interventions: Device: Moovcare® use

INTERVENTIONS:
Device: Moovcare® use — Moovcare® performs symptom monitoring by automatically delivering ePRO surveys on common symptoms experienced by lung cancer patients. Results are stored in a secure web-based portal for provider review. Providers will manage ePRO responses through a combination of reports graphically displaying responses over time and e-mail alerts about concerning levels or combinations of symptoms.

SUMMARY:
The purpose of this study is to demonstrate how Moovcare®, a mobile medical application, can be used to monitor Patient-Reported Outcomes (PROs) related to cancer treatment, cancer complications, and cancer relapse in patients with lung cancer. PROs are symptoms directly reported by patients through the completion of a survey. Up to 50 patients undergoing treatment and/or surveillance for new or existing diagnoses of lung cancer at the University of North Carolina's Lineberger Comprehensive Cancer Center will be prospectively enrolled to the use of the mobile medical application Moovcare® for 6 months. Moovcare® is not FDA approved, and its role in improving clinical care is being studied through this research. Moovcare® automatically delivers electronic patient reported outcome (ePRO) surveys on common symptoms experienced by lung cancer patients.

DETAILED DESCRIPTION:
This is a single site nonrandomized feasibility study of approximately 50 participants on treatment and/or surveillance for new or existing diagnoses of lung cancer who will be assigned to a single-arm involving monitoring of their patient-reported outcomes using a mobile medical application. The study procedures include monitoring of patient symptoms using automated weekly PRO surveys delivered by Moovcare® and assessment of outcomes including quality of life at baseline and at monthly intervals, as well as patient satisfaction at 6 months. The clinical care team will receive an alert if the PRO survey suggests increased or worsening symptoms. The care team will follow their usual protocols for the management of symptoms. The patient clinical information will also be abstracted from the medical record to assess clinical outcomes. The provider's satisfaction survey will be assessed via surveys.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Diagnosis of lung cancer (any histology, any stage) undergoing outpatient treatment and/or surveillance/monitoring at UNC.

   This may include stage I and II patients who have completed lung resection and/or are undergoing radiation, stage II and III patients receiving neoadjuvant, adjuvant, or definitive chemotherapy, stage IV patients undergoing active therapy or monitoring, patients undergoing surveillance for treated or untreated stage I-III lung cancer, and both limited and extensive small cell lung cancer. The study team will request the confirmation of the lung cancer diagnosis from the managing clinician. Patients can be enrolled at any point in their lung cancer treatment trajectory (i.e., not just at initiation of first-line treatment) after a diagnosis of lung cancer has been assigned by the treating clinician. This may include patients assigned a diagnosis of lung cancer without a tissue diagnosis.
3. Speaks and understands English
4. Reliable access to the internet and email
5. Access to a mobile phone (or device that can receive text messages for registration)

Exclusion Criteria:

1. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent or completing study procedures
2. Current participation in other PRO monitoring trials
3. Inability to read and speak English
4. Current incarceration

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gita Mody, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plans as of now to make IPD available to other researchers.

REFERENCES:
- [Derived] Stover AM, Deal AM, Medley CJ, Weiner AA, Novak L, Gentry AL, Hoch C, Weiss J, Pecot CV, Lee CB, O'Leary MC, Shrestha S, Chen H, Patel SA, Mody GN. Feasibility, Acceptability, and Utility of Remote Patient-Reported Outcomes Monitoring in Patients With Lung Cancer: A Moovcare(c) Study. Clin Lung Cancer. 2025 Dec;26(8):e660-e669.e1. doi: 10.1016/j.cllc.2025.07.016. Epub 2025 Aug 5. PMID 40850860
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 09/01/2021 through 03/14/2022 at one cancer center in North Carolina.
Pre-assignment Details: Forty-one participants started and completed the baseline assessment and thirty- three subjects completed the six-month assessment. Participant Flow and Baseline Characteristics are based on all participants who joined the study and completed baseline assessments.
Groups:
- Single-arm Moovcare®: Participants were assigned to the single-arm involving weekly monitoring of their patient-reported outcomes using Moovcare®.
  Moovcare® use: Moovcare® performs symptom monitoring by automatically delivering ePRO surveys on common symptoms experienced by lung cancer patients. Results are stored in a secure web-based portal for provider review. Providers will manage ePRO responses through a combination of reports graphically displaying responses over time and e-mail alerts about concerning levels or combinations of symptoms.
Period: Overall Study
Arm/Group | Single-arm Moovcare®
Started | 41
Completed (Forty-one participants completed the baseline assessment and thirty- three subjects completed the six-month evaluation.) | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects with lung cancer undergoing outpatient treatment and/or surveillance/monitoring and enrolled in the study and assessed per study criteria.
Groups:
- PRO Collected by Moovcare: Participants will be assigned to the single-arm involving weekly monitoring of their patient-reported outcomes using Moovcare®.
  Moovcare® use: Moovcare® performs symptom monitoring by automatically delivering ePRO surveys on common symptoms experienced by lung cancer patients. Results are stored in a secure web-based portal for provider review. Providers will manage ePRO responses through a combination of reports graphically displaying responses over time and e-mail alerts about concerning levels or combinations of symptoms.
Arm/Group | PRO Collected by Moovcare
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.51 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Self-reporting Symptoms Using Moovcare®
Description: Feasibility of self-reporting symptoms using Moovcare® is defined as the mean percentage of e-PRO surveys completed per subject using Moovcare® by 6 months or coming off study per protocol if sooner.
Time Frame: Up to 6 months
Population: Subjects enrolled in the study who started to use Moovcare and completed at least one survey questionnaire.
Measure: Mean (Standard Deviation); unit: percentage of e-PRO surveys completed
Arm/Group | Single-arm
Number analyzed (Participants) | 41
percentage of e-PRO surveys completed | 66.0 (34)

2. Secondary Outcome: Patient Satisfaction
Description: Percentage of subjects surveyed at 6 months in study satisfied with care team communication.
  Participant satisfaction was measured using a survey questionnaire that includes 11 mixed types of multiple-choice questions. Some questions have "yes" or "no" choices while others have multiple choices.
Time Frame: Baseline and at 6 months
Population: Subjects who are in the study and surveyed at 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Single-arm
Number analyzed (Participants) | 33
Participants | 30

3. Secondary Outcome: Health-related Quality of Life Change
Description: Health-related quality of life change was assessed using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) scores and the mean differences between 6 months and baseline was calculated.
  The EORTC QLQ-C30 is a cancer-specific instrument with 30 questions that incorporates 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social); 9 symptom scales (fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties); and a global health and quality-of-life scale. Most questions used 4 point scale (1 'Not at all' to 4 'Very much'); 2 questions used a 7-point scale (1 'Very poor' to 7 'Excellent'). The scores of these scales were averaged from the scores of the component items, transformed, and analyzed on a 0 - 100 scale. A higher score=better level of functioning or greater degree of symptoms.
Time Frame: Baseline and 6 months
Population: Subjects responded to EORTC QLQ-C30 both at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: Unite on a scale.
Arm/Group | Single-arm
Number analyzed (Participants) | 33
Unite on a scale. | -1.01 (21.32)

4. Secondary Outcome: Change in Health-related Quality of Life Lung Specific
Description: Health-related quality of life lung-specific change was assessed using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire and Lung Cancer Module (QLQ-LC13) scores and the mean differences between 6 months and baseline were calculated.
  EORTC QLQ-LC13 is a validated instrument to assess the quality of life and is composed of one multi-item scale. Possible scores range from 0 to 100; a higher score represents an increasing symptom level.
  A negative difference indicates quality of life improvement while a positive difference indicates worsened quality of life.
Time Frame: 6 months
Population: Subjects responded to EORTC QLQ-LC13 questionnaire at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: Unite on a scale.
Arm/Group | Single-arm
Number analyzed (Participants) | 33
Unite on a scale. | -1.01 (25.66)

5. Secondary Outcome: Participant Survey Completion Rate
Description: Percentage of participants who completed surveys completed at each weekly delivery time point using Moovcare.
Time Frame: Up to 6 months
Population: Subjects responded the questionnaire.
Measure: Number; unit: percentage of subjects
Arm/Group | Single-arm
Number analyzed (Participants) | 41
percentage of subjects
  Week 1 | 58.54
  Week 2 | 68.29
  Week 3 | 65.85
  Week 4 | 70.73
  Week 5 | 72.50
  Week 6 | 67.50
  Week 7 | 62.50
  Week 8 | 78.95
  Week 9 | 71.05
  Week 10 | 73.68
  Week 11 | 73.68
  Week 12 | 63.16
  Week 13 | 73.68
  Week 14 | 76.32
  Week 15 | 71.05
  Week 16 | 71.05
  Week 17 | 56.76
  Week 18 | 59.46
  Week 19 | 67.57
  Week 20 | 75.68
  Week 21 | 67.57
  Week 22 | 70.27
  Week 23 | 55.56
  Week 24 | 69.44
  Week 25 | 66.67

6. Secondary Outcome: Overall Survival
Description: Overall survival will be calculated using the Kaplan-Meier method, with time starting at enrollment and ending at last contact (6 months) or death, whichever came first.
Time Frame: From time of enrollment through last contact (Up to 6 months)
Population: Subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Single-arm
Number analyzed (Participants) | 41
Participants | 39

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Adverse events (AEs) are defined as any untoward or unexpected events or outcomes related to or possibly related to a subject's participation in the ePROs. AEs elicited in the free text portion of the ePRO survey. Any AEs and serious AEs will be reported to the UNC IRB using the IRB's web-based reporting system and per protocol. Serious AEs are not anticipated in patients related to undergoing the use of the ePRO survey system or participating in surveys for feedback on the ePRO system.
Arm/Group | Single-arm
All-Cause Mortality (participants affected / at risk) | 2/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT05011890/Prot_SAP_000.pdf